CLINICAL TRIAL: NCT05422495
Title: Effect of Playful Cognitive-motor Mobility Training on Balance, Gait and Cognition and on the Prevention of Falls in Seniors
Acronym: GATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-214
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Fall Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity (Experimental): cognitive-motor training : Cycléo device (COTTOS ®),
  Interventions: Behavioral: training with Cycléo device (COTTOS ®),
- No activity (Placebo Comparator): no training
  Interventions: Other: non intervention

INTERVENTIONS:
Behavioral: training with Cycléo device (COTTOS ®), — 8 weeks of training
  Arms: Activity
Other: non intervention — non intervention
  Arms: No activity

SUMMARY:
Falls in the elderly are the cause of considerable morbidity and mortality and constitute a public health problem with more than 9000 deaths in France among the over 65s following an accidental fall. Many scientific data suggest that regular physical activity has significant and long-lasting beneficial effects on the health of the elderly and is associated with better functional status, a lower risk of falls and improved cognitive functions. However, the attraction to physical activity fades over the years and the reasons mentioned by the elderly for a low practice of physical activity are multiple, the main one being the worsening of their state of health.

The objective of this study is therefore to evaluate the impact of playful, motivating mobility training, stimulating both mobility and cognition, for 8 weeks, on the balance and mobility of elderly people in EHPAD, in particular in conditions of dual-task well known to be at high risk of falling, as well as on the prevention of falls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged over 60, residing in nursing homes
* Subjects able to walk 15 meters unaided
* MMSE > 10
* Visual acuity in both eyes > 6/10
* Affiliated subject or beneficiary of a social security scheme
* Subject having given and signed an informed consent to participate in the study, or his/her guardian
* Subject having a sedentary activity or practicing a usual light to moderate physical activity (physical activities < 6 METs)

Exclusion Criteria:

* Subject with a parkinsonian syndrome, any impairment of the motor neuron, pain limiting the practice of physical activity
* Subject with a modification of less than 3 months of psychotropic drugs
* Subject practicing high intensity physical activity (> 6 METs)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-01-26 (Estimated); Study Completion 2024-01-26 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | change between baseline and 6 month
MMSE globale cognitive assesment | change between baseline and 6 month
Attention assessed by WAIS digit spans | change between baseline and 6 month
Executive functions assessed by the TMT A AND B | change between baseline and 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No